CLINICAL TRIAL: NCT06698978
Title: Interest of a Simplified Technique in Removable Complete Prosthesis Versus Conventional Technique in Edentulous Patients: a Multicenter Randomized Clinical Trial in Cross-over.
Brief Title: Simplified Technique in Removable Complete Prosthesis Versus Conventional Technique in Edentulous Patients
Acronym: IDEFIX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AOR22023
Record Dates: First submitted 2024-11-12; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Complete Edentulism
Keywords: removable prosthesis; simplified technique; cross-over; edentulous patients; conventional technique

STUDY DESIGN:
Intervention Model Description: The research consists of two 3-month treatment periods, spaced out by a 1-month wash-out period:
  Arm with complete removable denture according to the simplified protocol (PS) in period 1 (3 months), 1 month of wash-out then complete removable denture according to the conventional protocol (PC) in period 2 (3 months)
  Arm with complete removable denture according to the conventional protocol (PC) in period 1 (3 months), 1 month of wash-out then complete removable denture according to the simplified protocol (PS) in period 2 (3 months)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified(PS)/Conventional(PC) (Other): Complete removable denture according to the simplified protocol (PS) in period 1 (3 months), 1 month of wash-out then complete removable denture according to the conventional protocol (PC) in period 2 (3 months).
  Interventions: Other: Simplified protocol (PS)/Conventional protocol (PC)
- Conventional(PC)/Simplified (PS) (Other): Complete removable denture according to the conventional protocol (PC) in period 1 (3 months), 1 month of wash-out then complete removable denture according to the simplified protocol (PS) in period 2 (3 months).
  Interventions: Other: Conventional protocol (PC)/Simplified protocol (PS)

INTERVENTIONS:
Other: Simplified protocol (PS)/Conventional protocol (PC) — Complete removable denture according to the simplified protocol (PS) in period 1 (3 months), 1 month of wash-out then complete removable denture according to the conventional protocol (PC) in period 2 (3 months).
  Arms: Simplified(PS)/Conventional(PC)
Other: Conventional protocol (PC)/Simplified protocol (PS) — Complete removable denture according to the conventional protocol (PC) in period 1 (3 months), 1 month of wash-out then complete removable denture according to the simplified protocol (PS)in period 2 (3 months).
  Arms: Conventional(PC)/Simplified (PS)

SUMMARY:
This study compares a simplified complete removable denture technique (PS) to the conventional approach (PC) in edentulous patients. The goal is to demonstrate that the simplified technique is not inferior to the conventional method in terms of quality of life, measured by the OHIP-20 scale over three months. The trial also examines time, satisfaction, denture quality, cost, and masticatory performance.

Design:

This is a multicenter, randomized, cross-over study with 62 patients over 11 months of participation, including a one-month washout between treatments. Patients will receive both types of dentures, with the order randomized.

Population:

The trial targets edentulous patients, both uni- and bi-maxillary, aged 18 or older, with certain health and dental conditions.

Key Assessments:

Quality of Life: OHIP-20 scores are collected pre-treatment and after three months for each denture type.

Patient Satisfaction and Denture Quality: Assessed using modified Kapur criteria and patient satisfaction surveys.

Masticatory Performance: Evaluated with a chewing gum test. Medical Economic Impact: Cost analysis of each denture type.

Anticipated Outcomes:

Benefits include reducing costs and treatment times, enhancing accessibility to dentures, particularly for elderly and underserved populations, and adapting dental education to teach this simplified technique.

Centers Involved:

Seven centers across France, including AP-HP hospitals and private practices.

Timeline:

The inclusion period is 24 months, with a total study duration of 35 months.

DETAILED DESCRIPTION:
Despite the progress made in preventing caries and periodontal disease, edentury remains a major disability affecting function, nutrition, aesthetics and quality of life. In France, there were about two million edentulous in 2003 (HAS). It is estimated that the proportion of single-maxillary edentulous people in 65-74 years was 16.3% and 14.3% for bimaxillary edentulum. The population of complete edentulous is a fragile, often elderly population at risk of undernutrition and social isolation.

Since January 2021, the CCAM has imposed a RAC0 (remaining charge 0) for complete removable prostheses (PAC) with capped fees. These blocked fees make it difficult to produce high quality prostheses according to the conventional protocol. The blocked fees encourage liberal dentists to refer these patients to medical centres or hospital services. In addition, in areas of medical desertification, a shorter treatment time would be beneficial for patients and practitioners.

During the last five years, international literature has brought out simplified protocols to achieve PACs, shorter and more economical than conventional protocols. According to these studies there is no significant difference in quality of life for completely edentulous patients. However, these simplified AHRC implementation protocols are not harmonized and the simplification does not involve the same steps according to the protocols or the same classes of complete edentulous. In addition, these simplified protocols are not taught because they are too recent and with insufficient evidence from well-conducted clinical trials.

The hypothesis is that a new prosthetic realization technique with a single imprint, according to an innovative protocol, is not inferior in terms of quality of life than the conventional realization technique with two impressions in PAC.

The main objective of this study is to demonstrate the non-inferiority of a complete removable prosthesis made according to the simplified protocol compared to a complete removable prosthesis made according to the conventional protocol on quality of life, after 3 months of use of each prosthesis, in patients with complete single-maxillary or bi-maxillary edentesis (upper and/or lower arcada).

Primary Assessment Criterion : Variation in the total score on the OHIP-20 (Oral Health Impact Profile-20) questionnaire between inclusion and 3 months after prosthesis placement.

The OHIP 20 is a scale of oral quality of life, specific to total edentulousness, validated in French. It has 20 items rated from 1 to 6 (minimum score 20-maximum score 120). For each item, a score of 6 corresponds to an optimal quality of life.

Secondary objectives of research

* Compare the chair time between the two prostheses
* Compare patient satisfaction for each prosthesis using the Celebic & Knezovic-Zlataric questionnaire
* Compare the quality of prostheses using modified KAPUR criteria (retention and stability)
* Compare the cost of simplified restoration with that of conventional technique, estimate the national impact of the diffusion of simplified technique, and estimate the differential cost ratio results.
* Compare the patient's chewing performance between the two prostheses

Secondary evaluation criteria :

* Cumulative measurement of time spent (in minutes) at the chair for prosthesis fabrication and adjustment steps
* Measurement of patient satisfaction on different items for each prosthesis using the Celebic & Knezovic-Zlataric questionnaire at the beginning of each sequence and after 3 months of wearing each prosthesis
* Measurement of the quality of prostheses according to the Kapur score Modified (retention: 0 to 2; stability: 0 to 3)
* The full cost of manufacturing each prosthesis
* The additional cost per OHIP-20 point
* Measurement of masticatory performance after 3 months, for each prosthesis

Acts or Product being researched: Second PAC under the simplified protocol (PS)

This is a randomized, cross-over clinical trial consisting of two 3-month treatment periods spaced out by a 1-month wash-out period.

For complete bi-maxillary edentuses, a single arch is considered in the study but the other antagonist arch is performed according to a conventional protocol. The arcade considered will be randomized in case of bi-maxillary edentury and then randomization will be performed by minimization according to the following criteria: edentury arcade considered (maxillary or mandibular), center, complete edentury class (Grade 1-2 versus 3-4 according to the American College of Prosthodontists).

The cross-over test can be applied to complete edentulous disease as it is a chronic condition.

It should be noted that during the prosthetic realization stages, patients are carriers of their old removable prosthesis, possibly readapted.

A quality of life measurement (OHIP-20) will be performed with the old prosthesis before each of the prostheses (M4, M8) and 3 months after each of the PC or PS prostheses (M7, M11).

The time taken to complete each prosthesis will be measured in minutes from the imprint stage to the placement stage. In addition, the time spent on adjustments and focus will also be measured in minutes from the time of installation to 30 days after the insertion of new prostheses.

The patient will have to complete a specific satisfaction questionnaire using the Celebic & Knezovic-Zlataric questionnaire with the old prosthesis before wearing each of the prostheses (M4, M8) and 3 months after wearing each of the PC or PS prostheses (M7, M11).

The quality of the old prosthesis will be evaluated at PAC 1 to 4 months (M4) and the quality of each new prosthesis (PC or PS) after 3 months of wearing each of the prostheses (M7, M11). The quality of the prosthesis will be measured with the modified Kapur score: from 0 to 3 for retention and from 0 to 2 for stability, or an overall score of 0 to 5.

The chewing performance will be evaluated with the old prosthesis before wearing each of the prostheses (M4, M8) and 3 months after wearing each of the prostheses PC or PS (M7, M11). The chewing performance will be assessed using specific chewing gum. After 20 chewing cycles, we will collect the mixture of a two-coloured gum that is crushed in a calibrated way. The evaluation of the colour mix is evaluated with a grid that allows to assign a masticatory performance score on a scale from 1 to 5

At the end of the study, the patient chooses his or her preferred prosthesis. The other prosthesis is used as a back-up prosthesis.

Statistical analysis : The main analysis will be performed in the per-protocol (PP) and intent to treat (ITT) population. An interaction between effect period and treatment will be first sought; then, in the absence of interaction, the effect treatment will be analyzed. If an interaction is found, only the first period will be analyzed. Sensitivity analyses with adjustment to the initial quality of life level and adjustment to minimization criteria will also be performed.

The total OHIP-20 score at the end of each period will be compared between the two prostheses. The variation in OHIP-20 score will be expressed in each PC and PS prosthesis group by the mean standard deviation and the difference between the two prostheses will be calculated

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years
* Complete single-maxillary (upper or lower arcade) or bimaxillar (upper and lower arcade) edentesis paired with non-iatrogenic removable full dentures (possibly readapted)
* Edentulous arcade with healthy or sanitized mucosa
* Sufficient inter arcade space
* Free and informed consent
* Adequate understanding of written and spoken French
* Membership of a social security scheme

Exclusion Criteria:

* Patient unable to cooperate
* Presence of pathological lesions of the oral mucosa
* Parkinson's disease
* Gougerot-Sjögren's disease,
* Patient with cancer of the upper aerogribogastic tract
* Patient in psychiatric care
* Patient with neurological disease (vascular algia of the face, trigeminal neuralgia,...)
* Patient with xerostomia
* Allergy identified to resin
* Patient deprived of liberty by judicial or administrative decision
* Patient under legal protection (guardianship, curatorship)
* Patient under AME (State Medical Aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Variation in total OHIP-20 questionnaire score (Oral Health Impact Profile-20) between inclusion and 3 months after the prosthesis is inserted. | 3 months
  The OHIP 20 is a scale of oral quality of life, specific to total edentulousness, validated in French. It has 20 items rated from 1 to 6 (minimum score 20-maximum score 120). For each item, a score of 6 corresponds to an optimal quality of life.

SECONDARY OUTCOMES:
Compare the chair-based completion times between the two prostheses | up to 4 months
  Measurement of time spent (in minutes) at the chair for the stages of prosthesis construction and adjustment
Compare patient satisfaction for each prosthesis | 11 months
  Measurement of patient satisfaction on different items for each prosthesis using the Celebic and Knezovic-Zlataric questionnaire (Grade 1 to 5:Grade 1 Insufficient, Grade 2 Fair,Grade 3 Good, Grade 4 Very good, Grade 5 Excellent ) at the beginning of each sequence and after 3 months of wearing each prosthesis
Compare the quality of prostheses | 11 months
  Measurement of prosthesis quality according to the Kapur score Modified (retention: 0 to 2; stability: 0 to 3)
Compare the cost of simplified restoration with conventional technique, estimate the national impact of the diffusion of simplified technique and estimate the differential cost ratio results | 11 months
  compare the full cost of manufacturing each prosthesis
Masticatory performance between the two prostheses | 11 months
  Masticatory performance will be assessed with the old prosthesis before wearing each prosthesis (M4, M8) and 3 months after wearing each PC or PS prosthesis (M7, M11). Masticatory performance will be assessed using specific chewing gums. After 20 masticatory cycles, we will collect the mixture of a two-tone chewing-gum which is crushed in a calibrated manner.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe RIGNON-BRET, Study Director — APHP